### IDS BASELINE PARTICIPANTS' INFORMATION AND CONSENT SHEET

INTERVIEWER INSTRUCTION: Give this information sheet and the consent form to the respondent. Tell the respondent to read and understand both forms. Tell the respondent to ask you any questions about either form. If the respondent cannot read, then a witness should read the forms to the respondent.

### STUDY INFORMATION

| Study Title: Promoting Infant-Directed Speech (IDS) in Ghana |
|---|
| Hello. My name is I am a field officer from INNOVATIONS FOR POVERTY ACTION (IPA). I am talking with you today to conduct a research study: |
| Background of the Study |
| In this research study, we are interested in learning more about how children learn and how to improve |
| child education and child health. We hope this research will inform child education and health programs, |
| which may benefit this community and society. You were selected because you are visiting the |
| [insert name of Ghana Health Service clinic] for antenatal or postnatal care. We will be |
| surveying women between ages 18-40 visiting health facilities for antenatal and postnatal care for this |
| study. |
| <u>Procedures</u> |
| If you participate, trained surveyors from IPA will administer a questionnaire to you. These questions are |
| confidential, which means we will not tell anyone what you tell us. The questionnaires will cover |

If you participate, trained surveyors from IPA will administer a questionnaire to you. These questions are confidential, which means we will not tell anyone what you tell us. The questionnaires will cover household details, childcare, child health, and child education. We will not tell your family members, neighbors, or anyone else, so please answer as honestly as you can. If you don't want to answer a question, that is ok, but please answer if you can because it will help us a lot. To assure the accuracy of the survey data collection, we would like to record sections of this conversation. The recording will not be connected with your personal information and nobody outside the research team will have access to the recording. The recording will only be used by the research team to check accuracy. We will not record without your permission. If you do grant permission for this recording, you have the right to revoke recording permission at any time. This survey should take about 30 minutes to complete. We will ask to survey you again in-person sometime between August and September 2021.

### Confidentiality

All your responses will be anonymous / held in confidence. Only the researchers involved in this study and those responsible for research oversight will have access to the information you provide which identifies you or your child. Your responses will be numbered and the code linking the number with your names will be in a data file that can only be accessed through a secret password Researchers will keep your information secret/ confidential to the extent possible and allowable by the law. This project will be completed by December 2025 All records will be stored in a secure workspace until one year after that date. The records will then be destroyed.

## Risks and Benefits

The risks to participating in this study are inconvenience and loss of time. There are no direct benefits to you.

# Compensation

You will be offered a calendar as a thank you for participating in this study.

### Voluntary Participation

These surveys are voluntary. If you do not agree to participate or decide to end the survey later, there will be no penalty. Even if you agree to participate in the study, you won't have to answer all the requestions in the surveys if you don't want to. Also, even if you agree to participate in the study now, no one from IPA will be allowed to ask you additional questions in the future without asking for your consent again. As per the laid down national safety protocols during this COVID period to wear a nose

Form Has Been Approved by GHS - ERC for the Period 21 Jan, 2021 25 H. Jan, 2022 Sign... Pate Cond. Feb, 2921 Name. GHC-ERC Administrator

mask throughout the period of the questionnaire administration. If you decide to participate, we can provide you with a new nose mask you may keep after the interview.

# **Contact Information**

You can ask any questions that you have about the study now. If you later have a question about the study that you didn't think of now, you can contact:

-Innovations for Poverty Action 054-432-2614 (ask for Stephanie Adjovu, the senior research associate)

**Independent Contact:** If you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant, please contact:

- The Stanford Institutional Review Board (IRB) to speak to someone independent of the research team at (+001)650-723-2480 or toll free at +1-866-680-2906, or email at IRB2-Manager@lists.stanford.edu. You can also write to the Stanford IRB, Stanford University, 3000 El Camino Real, Five Palo Alto Square, 4th Floor, Palo Alto, CA 94306.
- The Ghana Health Service Ethics Review Committee at 050-353-9896 (ask for Nana Abena Kwaa Ansah Apatu) or email at ethics.research@ghsmail.org
- The Northwestern University Institutional Review Board may be contacted by phone at (312) 503-9338 or by email at irb@northwestern.edu

This is to Certify that this Study's Inform Conser'
Form Has Been Approved by GHS – ERC for the
Period 21 Date 26 Date 25 Sign.
Name GHC-ERC Administrator

## **CONSENT TO BE INTERVIEWED**

**Agreement to participate:** I have read the above information, or it has been read to me. I have had the opportunity to ask questions about it and any question I have asked has been answered to my satisfaction. I consent voluntarily to participate as subjects in this study and understand that I have the right to withdraw from the study at any time without it in any way affecting my further medical care.

| I agree to participate in this study Yes [] No [] I give permission for recording of my survey session. Yes [] No [] | | |
|---|---|---|
| Signature/Thumb print of Respondent | _ Date: | to the state of th |
| For Surveyors: I certify that the nature and purpose, the potential benefits with participating in this research have been explained to the above individual. | | associated |
| Signature of Surveyor: | Date: | |
| For Interpreter: I interpreted the purpose and contents of the Participants named participant to the best of my ability in [name of language, All questions, appropriate clarifications sort by the participant and answer his/her satisfaction. | to his proper unde | rstanding. |
| Signature of Interpreter: Contact | Date | : |
| For Witness: "I was present while the benefits, risks and procedures were questions were answered, and the volunteer has agreed to take part in the | | er. All |
| Signature of Witness (if necessary): | Date: | |

3